CLINICAL TRIAL: NCT07090772
Title: The Effectiveness of Different Therapeutic Jaw Position Determining Methods in Repositioning Splint Therapy for Temporomandibular Joint Disk Displacement Without Reduction：A Randomized Controlled Clinical Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Hao Yu, Director; Clinical Professor; dean of overseas education college; vice dean of school and hospital of stomatology, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025ECSS057
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Temporomandibular Disorder (TMD)
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- receive repositioning splint therapy with jaw position determined by mechanical articulator (Experimental): Participants will receive repositioning splint therapy with jaw position determined by mechanical articulator method for 3-6 months.
  Interventions: Procedure: Repositioning splint therapy with jaw position determined by mechanical articulator
- receive repositioning splint therapy with jaw position determined by ai-assisted virtual articulator (Experimental): Participants will receive repositioning splint therapy with jaw position determined by ai-assisted virtual articulator.
  Interventions: Procedure: Repositioning splint therapy with jaw position determined by ai-assisted virtual articulator
- receive repositioning splint therapy with jaw position determined by ai-assisted virtual patient (Experimental): Participants will receive repositioning splint therapy with jaw position determined by ai-assisted virtual patient
  Interventions: Procedure: Repositioning splint therapy with jaw position determined by ai-assisted virtual patient

INTERVENTIONS:
Procedure: Repositioning splint therapy with jaw position determined by mechanical articulator — The therapeutic jaw position will be determined by the following steps:
  1. Pre-treatment Jaw Position Recording Participants were seated upright with relaxed posture, eyes facing forward, and the Frankfort plane parallel to the floor. Intercuspal position (ICP) was recorded using silicone registration material. Edge-to-edge position of central incisors was recorded for protrusive position. Left/right lateral positions were recorded with opposing canines aligned.
  2. Transfer of Jaw Positions Following the manufacturer's protocol for the Artex CR mechanical facebow (Amann Girrbach, Austria) to transfer Participants' jaw positions.
  3. Determination of Therapeutic Position The Glenoid fossa was divided into 7 grids in the oblique-sagittal plane using Gelb's method, identifying grid 4 (Gelb 4/7) as the target condylar position.Condylar displacement knobs were set per VTO analysis.
  Incisal pin height was increased to establish vertical dimension.
  Arms: receive repositioning splint therapy with jaw position determined by mechanical articulator
Procedure: Repositioning splint therapy with jaw position determined by ai-assisted virtual articulator — The jaw position was determined by the following steps:
  1. AI-Based Segmentation and Reconstruction of Jaw Models CBCT DICOM data was imported into an ai-based craniomaxillofacial bone segmentation system to reconstruct 3D models of the jaws and dentition. The mandibular/maxillary bone models and dental arches were exported as .ply files. These .ply files were then imported into Exocad software.
  2. Virtual Transfer of Jaw Positions Bilateral AI-segmented medial pole points of the condyles and the right infraorbital point were annotated in cross-sectional views.A virtual articulator was added and registered to the facebow's reference planes and hinge axis. (3)Determination of Therapeutic Position Sagittal joint spaces (anterior/superior/posterior) were measured on cross-sectional views. The composite mandibular model was repositioned to the target occlusion using the "Move Mesh" function based on: Optimal mean joint space measurements and physiological condylar position.
  Arms: receive repositioning splint therapy with jaw position determined by ai-assisted virtual articulator
Procedure: Repositioning splint therapy with jaw position determined by ai-assisted virtual patient — The jaw position was determined by the following steps:
  1. AI-Based Segmentation and Reconstruction of Virtual Patients:
     CBCT DICOM data was imported into an ai-based craniomaxillofacial bone segmentation system to reconstruct 3D models of the jaws and dentition. The trajectory of mandibular movement was recorded by an electronic facebow.
  2. Virtual Transfer of Jaw Positions Bilateral AI-segmented medial pole points of the condyles and the right infraorbital point were annotated in cross-sectional views.A virtual articulator was added and registered to the facebow's reference planes and hinge axis. (3)Determination of Therapeutic Position Sagittal joint spaces (anterior/superior/posterior) were measured on cross-sectional views. The therapeutic position was determined based on: Optimal mean joint space measurements, physiological condylar position and optimal trajectory of mandibular movement.
  Arms: receive repositioning splint therapy with jaw position determined by ai-assisted virtual patient

SUMMARY:
The goal of this clinical trial is to learn if different therapeutic jaw position determining methods influence the efficacy of repositioning splint therapy for temporomandibular joint disk displacement without reduction. The main questions it aims to answer are:

Does different therapeutic jaw position determining methods influence the efficacy of repositioning splint therapy for temporomandibular joint disk displacement without reduction? Researchers will compare the efficacy of repositioning splint therapy made with different therapeutic jaw position determining methods for temporomandibular joint disk displacement without reduction.

Participants will:

Take repositioning splint made with different therapeutic jaw position determining methods every day for 3-6 months.

Visit the clinic once every 3 weeks for checkups and tests.

ELIGIBILITY:
Inclusion Criteria:

* Aged 13-50 years, with permanent dentition, possessing full autonomy in behavior and expression;
* Meeting the 2014 Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) diagnostic standards for irreducible temporomandibular joint disc displacement;
* MRI-confirmed unilateral irreducible disc displacement: At maximum intercuspation: Posterior band of disc located anterior to the 11:30 position, intermediate zone anterior to condyle; At maximum mouth opening: Intermediate zone remains anterior to condyle.

Exclusion Criteria:

* Systemic diseases, psychiatric disorders, or impaired consciousness;
* Pain-only disorders without articular pathology signs;
* Mandibular hypoplasia, TMJ tumors, or prior TMJ trauma;
* History of definitive TMJ disorder treatment.

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Condylar position as assessed by CBCT measurements | 3-6 months
  Condylar position of the three groups will be assessed after each treatment based on the measurements of sagittal joint spaces (anterior/superior/posterior) on CBCT's cross-sectional views.
Condylar repositioning rate as assessed by CBCT measurements | 3-6 months
  Using Mimics software, post-treatment condylar positions were analyzed and measured. The proportions of affected-side condyles reposition to the Gelb 4/7 position were compared across the three therapeutic jaw position determination methods.

SECONDARY OUTCOMES:
Fricton index as assessed by comprehensive physical examination to participants | 3-6 months
  Fricton index consists of dysfunction index and palpation index, which can quantify mandibular function and movement, palpation of muscles and other indicators, and is widely used to evaluate the clinical efficacy of temporomandibular disorders.
Dysfunction index as assessed by by comprehensive physical examination to participants | 3-6 months
  Dysfunction index refers to the comprehensive Index that reflect temporomandibular joint tenderness and functioning problems.
Palpation index as assessed by by comprehensive physical examination to participants | 3-6 months
  Palpation index refers to the comprehensive index that reflect muscle tenderness problems.

CONTACTS AND LOCATIONS:
Overall Officials: Hao Yu, PhD, MD, Principal Investigator — Fujian Medical University, China
Locations (1):
- Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No